CLINICAL TRIAL: NCT00820118
Title: ARNS 141 TIPI : A Pilot Trial to Assess the Ability of an Intermittent Antiretroviral Therapy in Maintaining an Immunological Stability in Antiretroviral naïve HIV Infected Adults, With CD4 Count Above 500/mm3
Brief Title: Early and Intermittent Antiretroviral Therapy in Naive HIV Infected Adults
Acronym: TIPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 141 TIPI
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: ANTIRETROVIRAL THERAPY; STRUCTURED TREATMENT INTERRUPTIONS; treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption; Atazanavir Sulfate; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intermittent treatment (Experimental): 6 months on antiretroviral treatment and 6 months off treatment
  Interventions: Drug: Structured treatment interruption

INTERVENTIONS:
Drug: Structured treatment interruption — The preferentially recommended treatment of the study is atazanavir boosted with ritonavir, associated with a fixed combination of abacavir and lamivudine or emtricitabine + tenofovir
  Usual dosage recommended :
  * atazanavir : 300 mg/d
  * ritonavir : 100 mg/d
  * abacavir 600 mg and lamivudine 300 mg : once a day
  * tenofovir 245 mg and emtricitabine 200 mg : once a day
  Other Names: Reyataz; Truvada; Kivexa; Treatment interruption; STI

SUMMARY:
The primary objective of the trial is to assess the ability of an early and intermittent antiretroviral therapy in maintaining an immunological stability in antiretroviral naive HIV infected adults, to offer a potential alternative strategy to differed and continuous antiretroviral treatment.This is a 2-year phase II, open-label, multicentric "proof of concept" trial. The patients included are treated following a pulse-therapy scheme, i.e. 6-month periods with once daily boosted-PI based therapy in alternance with 6-month periods without antiretroviral therapy. The preferentially recommended treatment of the study is atazanavir boosted with ritonavir, associated with a fixed combination of abacavir and lamivudine or emtricitabine + tenofovir.The patients are closely followed to assess the efficacy and the tolerance of the strategy, with clinical, biochemical, immunological, virological and pharmacokinetic evaluations.

ELIGIBILITY:
Inclusion Criteria:

* adult confirmed HIV-1 infection
* no previous treatment with antiretroviral drugs or interleukin-2
* CD4 count ≥ 500/mm3
* no active opportunistic infection
* written informed consent

Exclusion Criteria:

* non barrier contraception in women of child bearing potential, pregnant or breastfeeding woman, pregnancy project within the next 2 years
* HIV-2 infection (with or without HIV-1), recent HIV primary infection, resistance to trial drugs at study entry, Ag HBs+, HCV requiring specific therapy
* previous history of cerebrovascular accident or coronary heart disease, splenectomy
* previous CD4 count < 400/mm3
* CD4 percentage < 15%
* hemoglobin < 8 g/dl, neutrophils < 750/mm3, platelets < 100.000/mm3, creatinine clearance < 50 ml/mn, AST or ALT or total bilirubin > 3 ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
proportion of patients with mean CD4 count at M21 and M24 above or equal to the mean CD4 count at screening and inclusion, without experiencing a decrease below 400/mm3 throughout the study. | M21 and M24

SECONDARY OUTCOMES:
proportion of patients following the strategy of the trial and with AIDS related and non AIDS-related (cardiovascular, renal, hepatic, infectious, cancerous) serious clinical event | M12 and M24
number, type and time to AIDS and non AIDS-related serious clinical events | from week 0 to M24
number, type and time to clinical and biological events (whatever the grade of severity) | from week 0 to M24
existence and nature of HIV genotypic mutations associated with antiretroviral resistance | M9 and M24 and at any time visit in case of failure
proportion of patients having followed the strategy of the trial | from week 0 to M24
evolution of HIV RNA and HIV DNA throughout the study | from week 0 to M24 for RNA and each 6 months for DNA
Quality of life and observance (questionnaires) | QL each 6 months, observance at M1, M6, M13 and M18

CONTACTS AND LOCATIONS:
Overall Officials: Lionel PIROTH, MD, PHD, Principal Investigator — Hôpital de Dijon, France
Locations (1):
- Services maladies infectieuses et tropicales CHU, Dijon, France

REFERENCES:
- [Derived] Piroth L, Moinot L, Yeni P, Avettand-Fenoel V, Reynes J, Girard PM, Marchou B, Georget A, Rouzioux C, Autran B, Duvillard L, Chene G, Fagard C; ANRS 141 TIPI Trial Study Group. Immunity, inflammation and reservoir in patients at an early stage of HIV infection on intermittent ART (ANRS 141 TIPI Trial). J Antimicrob Chemother. 2016 Feb;71(2):490-6. doi: 10.1093/jac/dkv369. Epub 2015 Nov 14. PMID 26568566
- See also: Related Info — http://www.anrs.fr